CLINICAL TRIAL: NCT02783599
Title: A Phase 1b Trial to Assess the Modulation of Biological Markers in Patients With Potentially Resectable Soft Tissue Sarcoma Treated With Olaratumab Monotherapy Followed by Olaratumab Plus Doxorubicin Combination Therapy
Brief Title: A Study of Olaratumab (LY3012207) in Participants With Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15840; I5B-MC-JGDM (Other: Eli Lilly and Company); 2015-005018-31 (EudraCT Number)
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-02

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Olaratumab + Doxorubicin (Experimental): Cycle 1: Olaratumab 20 milligram per kilogram (mg/kg) given intravenously (IV) on Day 1 and Day 8 (21 day cycle).
  Cycle 2: Olaratumab 20 mg/kg given IV on Day 1 and Day 8 plus doxorubicin 75 mg/m2 given IV on Day 1 (21 day cycle).
  Cycle 3 through Cycle 7: Olaratumab 15 mg/kg given IV on Day 1 and Day 8 plus doxorubicin 75 mg/m2 given IV on Day 1 (21 day cycles).
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Olaratumab + Radiotherapy Addendum (Experimental): Olaratumab given IV on Day 1 and Day 8 (21 day cycle) concurrently with radiotherapy.
  Radiotherapy addendum was not implemented.
  Interventions: Drug: Olaratumab; Radiation: External Beam Radiotherapy

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207
Drug: Doxorubicin — Administered IV
  Arms: Olaratumab + Doxorubicin
Radiation: External Beam Radiotherapy
  Arms: Olaratumab + Radiotherapy Addendum

SUMMARY:
The purpose of this study is to evaluate potential biomarkers and method of action, efficacy and safety of olaratumab in participants with soft tissue sarcoma (STS).

ELIGIBILITY:
Inclusion Criteria:

* Have a histologically confirmed diagnosis of STS for which olaratumab and doxorubicin would be appropriate therapy. Participants with a diagnosis of Grade 1 liposarcoma are eligible if there is histological or radiographic evidence of evolution to more aggressive disease. Participants with Kaposi's sarcoma and gastrointestinal stromal tumors (GIST) will be excluded. Participants must have potentially resectable disease (as assessed by the study investigator) and have a primary tumor lesion deemed amenable to serial biopsy.
* For radiotherapy addendum only: Have a histologically confirmed diagnosis of STS of the extremities, Grade 2 or 3, >5 centimeters, for which olaratumab and radiotherapy would be appropriate therapy. Participants with Kaposi's sarcoma, GIST or myxoid liposarcoma will be excluded.
* Have consented to undergo mandatory serial peripheral whole blood and tumor tissue sampling.

Exclusion Criteria:

* Have active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis) at the time of enrollment. Participants with a history of a CNS metastasis previously treated with curative intent (for example, stereotactic radiation or surgery) that have not progressed on follow-up imaging, have been asymptomatic for at least 60 days and are not receiving systemic corticosteroids and or/anticonvulsants, are eligible. Participants with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before enrollment to rule out brain metastasis.
* Have received prior treatment with doxorubicin, epirubicin, idarubicin, and/or other anthracyclines or anthracenediones; the participant has received treatment with olaratumab or has participated in a prior olaratumab trial.
* For radiotherapy addendum only: Have received previous radiotherapy in the primary tumor lesion and/or prior treatment with olaratumab or has participated in a prior olaratumab trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (14):
- United States (9):
  - USC/Norris Comp Cancer Center, Los Angeles, California
  - Yale University School of Medicine, New Haven, Connecticut
  - All Children's Hospital, St. Petersburg, Florida
  - Moffitt Cancer Center & Research Inst, Tampa, Florida
  - Kansas City Cancer Center, Overland Park, Kansas
  - Washington University Medical Center, St Louis, Missouri
  - Levine Children's Hospital, Charlotte, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon, France
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan, Italy
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., London, United Kingdom

REFERENCES:
- See also: Click here for more information about this study: A Study of Olaratumab (LY3012207) in Participants With Soft Tissue Sarcoma — https://lillytrialguide.com/en/studies/soft-tissue%20sarcoma/JGDM#?postal=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are considered to have completed the study if they completed one cycle of monotherapy and all 6 cycles of combination therapy.
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered intravenously (IV) on Day 1 and Day 8 followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Period: Overall Study
Arm/Group | Olaratumab + Doxorubicin
Started | 51
Received At Least One Dose of Study Drug | 51
Completed | 11
Not Completed | 40
Not completed — Progressive disease | 23
Not completed — Surgical Resection | 10
Not completed — Adverse Event | 4
Not completed — Physician Decision | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered intravenously IV on Day 1 and Day 8, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17
  Italy | 3
  United Kingdom | 4
  France | 2
  Spain | 25
Circulating Tumor Cells (CTC) [Mean (Standard Deviation); unit: CTC per milliliter] — Population: All participants who received at least one dose of study drug and had evaluable blood samples for CTCs at baseline.
  CTC per milliliter
    Traditional CTC: number analyzed (Participants) | 35
    Traditional CTC | 2.183 (2.631)
    All Population CTC: number analyzed (Participants) | 35
    All Population CTC | 2.446 (2.797)
Platelet-Derived Growth Factor Receptor Alpha (PGDFRα ) and PGDFR Beta (β) [Mean (Standard Deviation); unit: relative gene expression units] — Population: All participants who received at least one dose of study drug and had evaluable tissue samples at baseline.
  relative gene expression units
    PGDFRα: number analyzed (Participants) | 37
    PGDFRα | 301.68 (570.79)
    PGDFRβ: number analyzed (Participants) | 37
    PGDFRβ | 812.49 (1260.23)
PDGF Canonical Ligands -A, -B, -C, -D [Mean (Standard Deviation); unit: relative gene expression units] — Population: All participants who received at least one dose of study drug and had evaluable tissue samples at baseline.
  relative gene expression units
    PGDF-A: number analyzed (Participants) | 37
    PGDF-A | 12.90 (18.46)
    PDGF-B: number analyzed (Participants) | 37
    PDGF-B | 230.62 (1151.87)
    PDGF-C: number analyzed (Participants) | 37
    PDGF-C | 227.68 (447.56)
    PDGF-D: number analyzed (Participants) | 37
    PDGF-D | 33.22 (69.99)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Enumeration of Circulating Tumor Cells (CTCs) in Whole Blood
Description: Enumeration of CTCs pre- and post- treatment with olaratumab may be a useful biomarker given the predilection for sarcomas to spread hematogenously.
Time Frame: Baseline, End of Cycle 1 (21 days)
Population: All participants who received one cycle of study drug and had evaluable blood samples for CTCs at baseline and post-olaratumab monotherapy.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Olaratumab: Olaratumab 20 mg/kg administered intravenously (IV) on Day 1 and Day 8 of Cycle 1.
Arm/Group | Olaratumab
Number analyzed (Participants) | 35
percent change
  Traditional CTCs | 846.93 (3260.60)
  All Population CTCs | 820.11 (3263.41)

2. Primary Outcome: Percent Change From Baseline in Gene Expression of Platelet-Derived Growth Factor Receptor Alpha (PGDFRα) and PGDFR Beta (β) in Tumor Tissue
Description: Over-activity of PDGF signaling is associated with the development of certain malignant diseases. Olaratumab is an IgG1 antagonist of PDGFRα.
Time Frame: Baseline, End of Cycle 1 (21 days)
Population: All participants who received at least one dose of study drug and had evaluable tissue samples at baseline and post-olaratumab monotherapy.
Measure: Mean (Standard Deviation); unit: percent change in gene expression
Groups:
- Olaratumab: Olaratumab 20 mg/kg administered IV on Day 1 and Day 8 of Cycle 1.
Arm/Group | Olaratumab
Number analyzed (Participants) | 37
percent change in gene expression
  PDGF Receptor α | 6162.86 (32383.49)
  PDGF Receptor β | 1246.25 (7024.82)

3. Primary Outcome: Percent Change From Baseline in Gene Expression of PDGF A, PDGF B, PDGF C, and PDGF-D Canonical Ligands in Tumor Tissue
Description: PDGF A, PDGF B, PDGF C, and PDGF D are platelet-derived growth factor canonical ligands associated with activation of PDGFR α and β.
Time Frame: Baseline, End of Cycle 1 (21 days)
Population: All participants who received at least one dose of study drug and had evaluable baseline tissue samples at baseline and post-olaratumab monotherapy.
Measure: Mean (Standard Deviation); unit: percent change in gene expression
Arm/Group | Olaratumab
Number analyzed (Participants) | 37
percent change in gene expression
  Canonical Ligand PDGF - A | 189.37 (672.91)
  Canonical Ligand PDGF - B | 602.01 (2798.92)
  Canonical Ligand PDGF - C | 1107.45 (6053.12)
  Canonical Ligand PDGF - D | 2630.36 (14425.92)

4. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression-free survival (PFS) is defined as the time from the date of first study dose to the first date of radiologic disease progression or death due to any cause. Progressive disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including the baseline sum if that is the smallest). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). The appearance of one or more new lesions is also considered progression.
Time Frame: Baseline to Objective Progression or Death from Any Cause (Up to 18 Months)
Population: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered intravenously (IV) on Day 1 and Day 8, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
months | 2.86 [1.41 to 9.72]

5. Secondary Outcome: Objective Response Rate (ORR): Percent of Participants With Best Overall Tumor Response of Complete Response (CR) or Partial Response (PR)
Description: Overall Response Rate (ORR) is defined as the percentage of participants achieving a best overall response of either Complete Response (CR) or Partial Response (PR) as determined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. CR is defined as a disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm and normalization of tumor marker results; PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters. The best overall response is the best response from the start of the treatment until progressive disease (PD)/recurrence.
Time Frame: Baseline to Measured Progressive Disease (Up to 18 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered IV on Day 1 and Day 8, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg olaratumab administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
percentage of participants | 11.8

6. Secondary Outcome: Disease Control Rate (DCR): Percent of Participants Who Exhibit Stable Disease (SD), CR or PR
Description: Disease control rate (DCR) is defined as the percentage of participants achieving a best overall response of CR, PR, or SD as determined by RECIST 1.1. CR is defined as a disappearance of all target lesions and any pathological lymph nodes must have reduction in short axis to <10 mm and normalization of tumor marker results; PR is defined as at least a 30% decrease in the sum of diameter of target lesions, taking as reference the baseline sum diameters; SD is defined as neither sufficient shrinking to qualify as PR nor sufficient increase to qualify for PD.
  Participants who do not have any post-baseline tumor response assessments for any reason are considered non-responders and are included in the denominator when calculating the response rate.
Time Frame: Baseline to Measured Progressive Disease (Up to 18 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered IV on Day 1 and Day 8, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
percentage of participants | 52.9

7. Secondary Outcome: Percentage of Participants With Resectable Tumors (Resectability Rate)
Description: Resectability rate is obtained when the total number of participants with resectable tumors is divided by the total number of participants. Resectability of a tumor is determined by the surgeon and multi-disciplinary team and dependent on tumor stage and the participants coexisting medical conditions.
Time Frame: Cycle 1 through Cycle 7 (Up to 6 Months)
Population: All participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 of Cycle 1, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3-7: olaratumab 15 mg/kg olaratumab administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
percentage of participants | 35.3 [22.4306 to 49.9318]

8. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Olaratumab Monotherapy
Description: Summary of Cmax of olaratumab monotherapy on Cycle 1 Day 1 and Day 8
Time Frame: Cycle 1 Days 1 and 8: Predose; 5 minutes(m) post-infusion
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- Olaratumab: Cycle 1: olaratumab 20 mg/kg administered IV on Day 1 and Day 8.
Arm/Group | Olaratumab
Number analyzed (Participants) | 51
micrograms per milliliter (µg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 47
  Cycle 1 Day 1 | 510 (22)
  Cycle 1 Day 8: number analyzed (Participants) | 45
  Cycle 1 Day 8 | 661 (24)

9. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Olaratumab
Description: Cmax of olaratumab Cycles 2 and 3 Day 1 and 8 of a 21-day cycle.
Time Frame: Cycle 2 Day 1: Predose, 5 minutes(m) post-infusion, 24 hours(h), 96h; Day 8:Predose, 5 m, and 24h, 48h, 96h, and 240h postdose; Cycle 3 Day 1 and Day 8: Predose and 5m post-infusion
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (µg/mL)
Groups:
- Olaratumab + Doxorubicin: Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
  Cycle 3: olaratumab 15 mg/kg administered IV on Day 1 and Day 8 and doxorubicin 75 mg/m2 IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
micrograms per milliliter (µg/mL)
  Cycle 2 Day 1: number analyzed (Participants) | 46
  Cycle 2 Day 1 | 624 (26)
  Cycle 2 Day 8: number analyzed (Participants) | 42
  Cycle 2 Day 8 | 711 (28)
  Cycle 3 Day 1: number analyzed (Participants) | 29
  Cycle 3 Day 1 | 521 (30)
  Cycle 3 Day 8: number analyzed (Participants) | 28
  Cycle 3 Day 8 | 601 (32)

10. Secondary Outcome: Number of Participants With Anti-Olaratumab Antibodies
Description: A participant is counted as positive if they had at least one anti-olaratumab antibody positive result during the study.
Time Frame: Predose Cycle 1 Day 1 through Follow-Up (Up to 8 Months)
Population: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Olaratumab + Doxorubicin
Number analyzed (Participants) | 51
Participants | 1

ADVERSE EVENTS:
Time Frame: Baseline to end of study (Up to 46 months)
Description: All participants who received at least one dose of study drug.
Groups:
- Olaratumab + Doxorubicin: Cycle 1: olaratumab 20 mg/kg administered intravenously (IV) on Day 1 and Day 8, followed by up to 6 cycles (Cycle 2 - Cycle 7) of combination therapy with olaratumab and doxorubicin.
  Cycle 2: olaratumab 20 mg/kg administered IV on Day 1 and Day 8 and 75 mg/m2 of doxorubicin IV on Day 1.
  Cycle 3-7: olaratumab15mg/kg administered IV on Day 1 and Day 8 and 75 mg/m2 of doxorubicin IV on Day 1.
Arm/Group | Olaratumab + Doxorubicin
All-Cause Mortality (participants affected / at risk) | 3/51
Serious Adverse Events (participants affected / at risk) | 22/51
Other Adverse Events (participants affected / at risk) | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Doxorubicin (N=51)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (11)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olaratumab + Doxorubicin (N=51)
Anaemia (Blood and lymphatic system disorders) | 11 (22)
Neutropenia (Blood and lymphatic system disorders) | 10 (15)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 5 (7)
Constipation (Gastrointestinal disorders) | 20 (27)
Diarrhoea (Gastrointestinal disorders) | 12 (17)
Dyspepsia (Gastrointestinal disorders) | 6 (8)
Flatulence (Gastrointestinal disorders) | 4 (5)
Nausea (Gastrointestinal disorders) | 27 (48)
Stomatitis (Gastrointestinal disorders) | 22 (33)
Vomiting (Gastrointestinal disorders) | 12 (14)
Asthenia (General disorders) | 13 (30)
Chills (General disorders) | 4 (4)
Fatigue (General disorders) | 24 (38)
Oedema peripheral (General disorders) | 7 (8)
Pyrexia (General disorders) | 9 (13)
Urinary tract infection (Infections and infestations) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (7)
Procedural pain (Injury, poisoning and procedural complications) | 4 (5)
Blood creatinine increased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 11 (17)
Platelet count decreased (Investigations) | 4 (7)
White blood cell count decreased (Investigations) | 9 (13)
Decreased appetite (Metabolism and nutrition disorders) | 17 (21)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Dizziness (Nervous system disorders) | 9 (11)
Dysgeusia (Nervous system disorders) | 6 (8)
Headache (Nervous system disorders) | 8 (9)
Anxiety (Psychiatric disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (8)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 16 (17)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
Radiotherapy addendum was not implemented due to business decisions. There were no safety or efficacy issues related to the addendum that contributed to this decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT02783599/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT02783599/SAP_001.pdf